CLINICAL TRIAL: NCT01527292
Title: Randomized Phase II Trial of Stereotactic Radiation Therapy (SRT) Versus SRT Plus Vertebral Augmentation Procedure (VAP) for Vertebral Metastasis
Brief Title: Phase II Trial of Stereotactic Radiation Therapy (SRT) Versus SRT Plus Vertebral Augmentation Procedure (VAP) for Vertebral Metastasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Shiao Yuo Woo, Chair-Radiation Oncology, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCC-RAD-11-01
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2016-01

CONDITIONS: Vertebral Metastasis
Keywords: Vertebral Metastasis; pain control; VAP; SRT+VAP
MeSH Terms: conditions — Agnosia | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Baseline Assessments and followup assessments are the same for both arms. Control group Intervention: Stereotactic Radiation Therapy only
  Interventions: Radiation: Stereotactic Radiation Therapy
- Treatment Group (Experimental): SRT with Vertebral Augmentation Procedure Baseline Assessments and followup assessments are the same for both arms. Treatment group Intervention: Stereotactic Radiation Therapy with Vertebral Augmentation Procedure
  Interventions: Radiation: SRT with Vertebral Augmentation Procedure

INTERVENTIONS:
Radiation: Stereotactic Radiation Therapy — SRT only
  Other Names: Stereotactic Radiosurgery
  Arms: Control Group
Radiation: SRT with Vertebral Augmentation Procedure — SRT with VAP
  Other Names: Stereotactic Radiosurgery with VAP
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to determine pain control rate (Percentage of patients in each arm that achieve pain control) at the treated site(s) at 1 month, 2-4 months and 5-6 months post-treatment.

DETAILED DESCRIPTION:
Eligible Vertebral Metastatic Lesion/s-> randomized-> SRT versus SRT+ VAP Stereotactic Radiation Therapy(SRT): 16 Gy X 1 Evaluation: prior to treatment; 1 month, 2-4 months, 5-6 months and 1 year post-treatment

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. ECOG performance status 0-1.
3. Known histologically proven malignancy.
4. Localized osteolytic spine metastases from T7 to L5 demonstrated by MRI, CT, PET or bone scan: a solitary spine metastasis; two separate spine levels; or up to 3 separate sites (each site may have a maximal involvement of 2 contiguous vertebral bodies with or without a paraspinal mass of no more than 5 cm).
5. Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential.
6. Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control.
7. Numerical Rating Pain Scale (NRPS) and movement-related pain score(MRPS) within two (2) weeks prior to registration.
8. The patient must have a score of ≥ 5 for at least one of the planned sites for SRT.
9. Patients must provide study specific informed consent prior to study entry.
10. Required Pre-treatment Evaluations: baseline Numerical Rating Pain Scale (NRPS), movement-related pain score, dose and frequency of all pain medications; QOL Measure using the Oswestry Disability Questionnaire, and EuroQOL(EQ-5D).

Exclusion Criteria:

1. Non-ambulatory patients.
2. Frank spinal cord compression or epidural compression within 3 mm of the spinal cord.
3. Osteoblastic vertebral metastasis.
4. Prior radiation to the index spine.
5. Patients with rapid neurologic decline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-05-02 (Actual); Study Completion 2015-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shiao Y Woo, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Baseline Assessments and followup assessments are the same for both arms. Treatment group Intervention: Stereotactic Radiation Therapy with Vertebral Augmentation Procedure
  SRT with Vertebral Augmentation Procedure: SRT with VAP
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 0 | 3
Completed | 0 | 0
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Population: Trial did not meet enrollment goal. Investigator did not analyze data due to low enrollment and early termination of trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 61 [56 to 64] | 61 [56 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 3
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Pain Scale (NRPS) Change in Patients
Description: To determine pain control rate (Percentage of patients in each arm that achieve pain control) at the treated site(s)at 1 month, 2-4 months and 5-6 months post-treatment and to validate of the movement-related pain score
Time Frame: For 6 months post treatment
Population: Data not analyzed due to low enrollment and early termination of study
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Reduction of Pain Estimate
Description: To estimate the relative quantitative reduction of pain from baseline in patients in each arm.
Time Frame: For 1 year post treatment
Population: Data not analyzed due to low enrollment and early termination of study
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life Estimate
Description: To estimate the quality of life using the Oswestry Disability Questionnaire
Time Frame: For 1 year post treatment
Population: Data not analyzed due to low enrollment and early termination of study
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Feasibility Rate Estimation
Description: To estimate the feasibility rate of the study procedure (the percentage of patients in overall and each arm that complete the treatment).
Time Frame: For 1 year post treatment
Population: Data not analyzed due to low enrollment and early termination of study
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Toxicity Rate Estimation
Description: To estimate the toxicities of the treatment
Time Frame: For 1 year post treatment
Population: Data not analyzed due to low enrollment and early termination of study
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Vertebra Measurement
Description: To measure the dimensions of the treated vertebra(e) at 1 year
Time Frame: For 1 year post treatment
Population: Data not analyzed due to low enrollment and early termination of study
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes